CLINICAL TRIAL: NCT02978781
Title: A Phase 2a, Double-Blind, Placebo-Controlled, Randomized Withdrawal Study Evaluating the Efficacy, Safety, Tolerability, and Pharmacokinetics of SAGE-217 in the Treatment of Subjects With Essential Tremor
Brief Title: A Study to Evaluate SAGE-217 in Participants With Essential Tremor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 217-ETD-201
Record Dates: First submitted 2016-10-24; First posted 2016-12-01 (Estimated); Results first posted 2021-02-17 (Actual); Last update posted 2023-11-28 (Actual); Status verified 2023-11

CONDITIONS: Essential Tremor
Keywords: Tremor
MeSH Terms: conditions — Essential Tremor; Tremor | interventions — zuranolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A: SAGE-217 Oral Solution (Experimental): Participants received SAGE-217 10 mg oral solution on Day 1, 20 mg on Day 2 and 30 mg on Days 3 to 7 with food in the morning.
  Interventions: Drug: SAGE-217
- Part A: SAGE-217 Capsules (Experimental): Participants received SAGE-217 10 mg capsules on Day 1, 20 mg on Day 2 and 30 mg on Days 3 to 7, orally, with food in the morning.
  Interventions: Drug: SAGE-217
- Part B: Placebo (Placebo Comparator): Participants who received maximum tolerated dose of SAGE-217 in Part A and achieved response on Day 8 were randomized to receive to SAGE-217 matching placebo for 7 days beginning on Day 8 with food in the morning.
  Interventions: Drug: Placebo
- Part B: SAGE-217 Capsules (Experimental): Participants who received maximum tolerated dose of SAGE-217 in Part A and achieved response on Day 8 were randomized to receive to SAGE-217 for 7 days beginning on Day 8 with food in the morning.
  Interventions: Drug: SAGE-217
- Part C: SAGE-217 Capsules (Experimental): Participants received SAGE-217 10 mg capsules on Day 1, 20 mg on Day 2, 30 mg on Day 3, orally, with food in the evening. Beginning on Day 4 through Day 14, participants received a 40-mg total daily dose (administered as 10 mg with food in the morning and 30 mg with food in the evening).
  Interventions: Drug: SAGE-217

INTERVENTIONS:
Drug: SAGE-217 — SAGE-217 Oral Solution
  Arms: Part A: SAGE-217 Oral Solution
Drug: SAGE-217 — SAGE-217 Capsules
  Arms: Part A: SAGE-217 Capsules; Part B: SAGE-217 Capsules; Part C: SAGE-217 Capsules
Drug: Placebo — SAGE-217 matching placebo capsules
  Arms: Part B: Placebo

SUMMARY:
This study is a three-part, multicenter, Phase 2a study to evaluate the efficacy, safety, tolerability, and pharmacokinetics of SAGE-217 in adult participants with essential tremor.

DETAILED DESCRIPTION:
Part A of the study was an open-label design with morning dosing of SAGE-217 for 7 days and included 16 participants, 8 of whom qualified for, and entered, Part B.

Part B had a double-blind, placebo-controlled, randomized withdrawal design with morning dosing for 7 days.

Part C was an open-label design with morning and evening dosing for 14 days and included a different set of 18 participants.

Parts A and B were stopped early (in advance of the planned sample size).

This study was previously posted by Sage Therapeutics. In November 2023, sponsorship of the trial was transferred to Biogen.

ELIGIBILITY:
Key Inclusion Criteria:

* Participant must have a diagnosis of Essential Tremor (ET), defined as bilateral postural tremor and kinetic tremor, involving hands and forearms, that is visible and persistent and the duration is >5 years prior to screening.

Key Exclusion Criteria:

* Participant has presence of abnormal neurological signs other than tremor or Froment's sign.
* Participant has presence of known causes of enhanced physiological tremor.
* Participant has concurrent or recent exposure (14 days prior to admission visit) to tremorogenic drugs.
* Participant has had direct or indirect trauma to the nervous system within 3 months before the onset of tremor.
* Participant has historical or clinical evidence of tremor with psychogenic origin.
* Participant has convincing evidence of sudden tremor onset or evidence of stepwise deterioration of tremor.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2017-03-24 (Actual); Primary Completion 2017-11-22 (Actual); Study Completion 2017-12-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (26):
- United States (26):
  - Sage Investigational Site, Anniston, Alabama
  - Sage Investigational Site, Little Rock, Arkansas
  - Sage Investigational Site, Rogers, Arkansas
  - Sage Investigational Site, Cerritos, California
  - Sage Investigational Site, Fountain Valley, California
  - Sage Investigational Site, Oceanside, California
  - Sage Investigational Site, San Diego, California
  - Sage Investigational Site, Englewood, Colorado
  - Sage Investigational Site, Clearwater, Florida
  - Sage Investigational Site, DeLand, Florida
  - Sage Investigational Site, Lauderdale Lakes, Florida
  - Sage Investigational Site, Orlando, Florida
  - Sage Investigational Site, Ormond Beach, Florida
  - Sage Investigational Site, St. Petersburg, Florida
  - Sage Investigational Site, Tampa, Florida
  - Sage Investigational Site, Atlanta, Georgia
  - Sage Investigational Site, Decatur, Georgia
  - Sage Investigational Site, Chicago, Illinois
  - Sage Investigational Site, Urbana, Illinois
  - Sage Investigational Site, Springfield, Missouri
  - Sage Investigational Site, St Louis, Missouri
  - Sage Investigational Site, Raleigh, North Carolina
  - Sage Investigational Site, Cincinnati, Ohio
  - Sage Investigational Site, Dayton, Ohio
  - Sage Investigational Site, Nashville, Tennessee
  - Sage Investigational Site, Fort Worth, Texas

IPD SHARING:
Plan to Share IPD: Yes
In accordance with Biogen's Clinical Trial Transparency and Data Sharing Policy on https://www.biogentrialtransparency.com/
URL: https://vivli.org/

REFERENCES:
- See also: Related Info — http://www.sagerx.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 34 participants were enrolled in the study from 11 investigation sites in United States.
Pre-assignment Details: A total of 34 participants enrolled in the study. 16 participants received either SAGE-217 oral solution (N=2) or capsules (N=14) in Part A; 8 participants who tolerated a dose ≥10 mg in Part A and achieved response on Day 8 were randomized (1:1) in Part B to Placebo or SAGE-217 capsules.18 participants received SAGE-217 capsules in Part C.
Groups:
- Part B: Placebo: Participants who tolerated a ≥10 mg dose of SAGE-217 in Part A and achieved response (≥30% reduction in kinetic tremor) on Day 8 were randomized to receive SAGE-217 matching placebo for 7 days beginning on Day 8 with food in the morning. Participants received placebo capsules to match their maximum tolerated SAGE-217 dose as determined in Part A.
- Part B: SAGE-217 Capsules: Participants who tolerated a ≥10 mg dose of SAGE-217 in Part A and achieved response on Day 8 were randomized to receive maximum tolerated SAGE-217 in Part A for 7 days beginning on Day 8 with food in the morning. Participants received their maximum tolerated SAGE-217 dose as determined in Part A.
Period: Part A
Arm/Group | Part A: SAGE-217 Oral Solution | Part A: SAGE-217 Capsules | Part B: Placebo | Part B: SAGE-217 Capsules | Part C: SAGE-217 Capsules
Started | 2 | 14 | 0 | 0 | 0
Completed | 1 | 12 | 0 | 0 | 0
Not Completed | 1 | 2 | 0 | 0 | 0
Not completed — Adverse Event | 1 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Period: Part B
Arm/Group | Part A: SAGE-217 Oral Solution | Part A: SAGE-217 Capsules | Part B: Placebo | Part B: SAGE-217 Capsules | Part C: SAGE-217 Capsules
Started | 0 | 0 | 4 (Include participants who tolerated a dose ≥10 mg in Part A and achieved response on Day 8.) | 4 (Include participants who tolerated a dose ≥10 mg in Part A and achieved response on Day 8.) | 0
Completed | 0 | 0 | 4 | 3 | 0
Not Completed | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 1 | 0
Period: Part C
Arm/Group | Part A: SAGE-217 Oral Solution | Part A: SAGE-217 Capsules | Part B: Placebo | Part B: SAGE-217 Capsules | Part C: SAGE-217 Capsules
Started | 0 | 0 | 0 | 0 | 18
Completed | 0 | 0 | 0 | 0 | 14
Not Completed | 0 | 0 | 0 | 0 | 4
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 1
Not completed — Tremor not improved due to Topamax discontinuation | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The safety population included participants who received at least one dose of study drug in Part A and Part C. Participants who were randomized in Part B are not displayed here, as they are the same participants who tolerated study drug and were in the safety population for Part A. Part B participants are captured in the efficacy population.
Groups:
- Part A: SAGE-217 Oral Solution: Participants received SAGE-217 10 mg on Day 1, 20 mg on Day 2 and 30 mg daily on Days 3 to 7 as an oral solution with food in the morning.
- Part A: SAGE-217 Capsules: Participants received a 10-mg dose of SAGE-217, capsules administered with food in the morning on Day 1, 20 mg with food on Day 2 and 30 mg with food daily on Days 3 to 7.
- Part C: SAGE-217 Capsules: Participants received a 10-mg dose of SAGE-217 administered with food in the evening on Day 1, 20 mg with food in the evening on Day 2, and 30 mg with food in the evening on Day 3. From From Day 4 through 14 participants received a total 40-mg daily dose with food in the evening.
- Total: Total of all reporting groups
Arm/Group | Part A: SAGE-217 Oral Solution | Part A: SAGE-217 Capsules | Part C: SAGE-217 Capsules | Total
Number analyzed (Participants) | 2 | 14 | 18 | 34
Age, Continuous [Mean (Standard Deviation); unit: years] | 71.5 (0.71) | 62.4 (8.34) | 65.8 (8.21) | 64.7 (8.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 7 | 10 | 18
  Male | 1 | 7 | 8 | 16
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Black or African American | 1 | 3 | 0 | 4
  White | 1 | 11 | 18 | 30
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Not Hispanic or Latino | 2 | 14 | 18 | 34
Region of Enrollment [Number; unit: participants]
  United States | 2 | 14 | 18 | 34

OUTCOME MEASURES:

1. Primary Outcome: Part A: Change From Baseline in Accelerometer-based Kinesia Kinetic Tremor Combined Score at Day 7
Description: The accelerometer-based Kinesia kinetic tremor combined score is the sum of Kinesia kinetic tremor scores across both sides of the body. Tremor is measured using a motion sensor that transmits raw data to a computer where it converts the tremor amplitude to a Kinesia score of 0 to 4 based on validated algorithms; the total score ranges from 0 to 8, higher scores indicate more severe tremor. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) and Day 7 (8 hours postdose)
Population: Efficacy population (Part A; capsules) included all participants who received at least 1 dose of SAGE-217 capsule formulation in Part A and had at least 1 postdose efficacy evaluation. Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: SAGE-217 Capsules
Number analyzed (Participants) | 14
score on a scale
  Baseline (Day 1) | 4.36 (1.199)
  Change from Baseline at Day 7 (8 hours postdose): number analyzed (Participants) | 12
  Change from Baseline at Day 7 (8 hours postdose) | -0.69 (1.115)

2. Primary Outcome: Part B: Change From Randomization in Accelerometer-based Kinesia Kinetic Tremor Combined Score at Day 14
Description: The accelerometer-based Kinesia kinetic tremor combined score is the sum of Kinesia kinetic tremor scores across both sides of the body. Tremor is measured using a motion sensor that transmits raw data to a computer where it converts the tremor amplitude to a Kinesia score of 0 to 4 based on validated algorithms; the total score ranges from 0 to 8, higher scores indicate more severe tremor. A negative change from Randomization indicates improvement.
Time Frame: Randomization (Day 8, predose) and Day 14 (predose)
Population: The Efficacy Population included all participants who completed at least one dose of study drug in Part B and had at least one post-randomization efficacy evaluation.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Part B: Placebo: Participants who tolerated a ≥10 mg dose of SAGE-217 in Part A and achieved response on Day 8 were randomized to receive SAGE-217 matching placebo for 7 days beginning on Day 8 with food in the morning. Participants received placebo capsules to match their maximum tolerated SAGE-217 dose as determined in Part A.
- Part B: SAGE-217 Capsules: Participants who tolerated a ≥10 mg dose of SAGE-217 in Part A and achieved response on Day 8 were randomized to receive SAGE-217 for 7 days beginning on Day 8 with food in the morning. Participants received their maximum tolerated SAGE-217 dose as determined in Part A.
Arm/Group | Part B: Placebo | Part B: SAGE-217 Capsules
Number analyzed (Participants) | 4 | 4
score on a scale
  Randomization (Day 8) | 3.33 (0.714) | 4.13 (1.438)
  Change from Randomization at Day 14 (predose) | 0.20 (0.271) | 0.15 (0.191)
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: SAGE-217 Capsules; Change from Randomization at Day 14 (predose); Test type: Superiority; p = 0.9143, Mixed Model for Repeated Measures (MMRM); Least Squares Mean Difference = 0.02, 95% CI 2-sided [-0.44 to 0.49], Standard Error of Mean 0.227 — Least squares mean difference from Randomization (SAGE-217 - placebo); MMRM model was used for analysis with change from randomization of the Kinesia kinetic tremor combined scores as the dependent variable, treatment group by study visit/time point interaction as fixed effects, and randomization value as a covariate

3. Primary Outcome: Part C: Change From Baseline in the Accelerometer-based Kinesia Upper Limb Tremor Combined Score at Day 15
Description: The accelerometer-based Kinesia upper limb total score is the sum of the individual item scores across both sides of the body. The individual items included forward outstretched postural tremor (FOPT), lateral "wing beating" postural tremor (LWBPT), and kinetic tremor (KT) scores from both sides of the body. Each upper limb individual item question score for each side of the body ranges from 0 to 4. The Kinesia upper limb total score ranges from 0 to 24, with higher scores indicating more tremors/greater tremor amplitude. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) and Day 15
Population: The Efficacy Population consisted of all participants who completed at least 1 dose of study drug in Part C and had at least 1 postdose efficacy evaluation. Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part C: SAGE-217 Capsules
Number analyzed (Participants) | 16
score on a scale
  Baseline (Day 1) | 11.68 (3.822)
  Change from Baseline at Day 15: number analyzed (Participants) | 12
  Change from Baseline at Day 15 | -2.22 (2.956)
Statistical Analysis 1: Comparison: Part C: SAGE-217 Capsules; Change from Baseline at Day 15; Test type: Other; p = 0.0529, Mixed Model for Repeated Measures (MMRM); Least Squares Mean Difference = -1.74, 95% CI 2-sided [-3.50 to 0.03], Standard Error of Mean 0.815 — Least squares mean difference from Baseline (SAGE-217); [other analysis details as in outcome 2, analysis 1]

4. Secondary Outcome: Part A: Change From Baseline in Kinesia Upper Limb Total Score at Day 7
Description: The accelerometer-based Kinesia upper limb total score is the sum of Kinesia kinetic tremor scores across both sides of the body. The individual items included forward outstretched postural tremor (FOPT), lateral "wing beating" postural tremor (LWBPT), and kinetic tremor (KT) scores from both sides of the body. Each upper limb individual item question score for each side of the body ranges from 0 to 4. The Kinesia upper limb total score ranges from 0 to 24, with higher scores indicating more tremors/greater tremor amplitude. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) and Day 7 (8 hours postdose)
Population: Efficacy population (Part A; capsules) included all participants who received at least 1 dose of SAGE-217 capsule formulation in Part A and had at least 1 postdose efficacy evaluation. Number analyzed is the number of participants with data available for analysis at the given timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: SAGE-217 Capsules
Number analyzed (Participants) | 14
score on a scale
  Baseline (Day 1) | 10.50 (4.395)
  Change from Baseline at Day 7 (8 hours postdose): number analyzed (Participants) | 12
  Change from Baseline at Day 7 (8 hours postdose) | -2.40 (3.395)

5. Secondary Outcome: Part A: Change From Baseline in Kinesia Upper Limb Individual Item Score at Day 7
Description: The accelerometer-based Kinesia upper limb total score is the sum of Kinesia kinetic tremor scores across both sides of the body. The individual items included forward outstretched postural tremor (FOPT), lateral "wing beating" postural tremor (LWBPT), and kinetic tremor (KT) scores from both sides of the body. Each upper limb individual item question score for each side of the body ranges from 0 to 4, with higher scores indicating more tremors/greater tremor amplitude. The Kinesia upper limb total score ranges from 0 to 24, with higher scores indicating more tremors/greater tremor amplitude. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) and Day 7 (8 hours [hr] postdose [pd])
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: SAGE-217 Capsules
Number analyzed (Participants) | 14
score on a scale
  FOPT at Baseline (Day 1) | 2.51 (1.749)
  Change from Baseline in FOPT at Day 7 (8 hr pd): number analyzed (Participants) | 12
  Change from Baseline in FOPT at Day 7 (8 hr pd) | -0.74 (1.339)
  LWBPT at Baseline (Day 1) | 3.63 (1.695)
  Change from Baseline in LWBPT at Day 7 (8 hr pd): number analyzed (Participants) | 12
  Change from Baseline in LWBPT at Day 7 (8 hr pd) | -0.97 (1.312)
  Kinetic tremor at Baseline (Day 1) | 4.36 (1.199)

6. Secondary Outcome: Part A: Change From Baseline in the Tremor Research Group (TRG) Essential Tremor Rating Assessment Scale (TETRAS) Upper Limb Total Score at Day 7
Description: The TETRAS performance subscale upper limb total score is the sum of the TETRAS individual item scores from both sides of the body. The TETRAS individual item score included TETRAS Performance Subscale item 4a, 4b and 4c scores [4a: forward outstretched postural tremor (FOPT) and 4b: lateral "wing beating" postural tremor (LWBPT) scores and 4c: Kinetic tremor (KT) score] from both sides of the body. Each individual item score ranges from 0 to 4; The total upper limb score ranges from 0 to 24, higher scores indicate more severe tremor. A negative change indicates improvement.
Time Frame: Baseline (Day 1) and Day 7 (8 hours postdose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: SAGE-217 Capsules
Number analyzed (Participants) | 14
score on a scale
  Baseline (Day 1) | 12.86 (2.373)
  Change from Baseline at Day 7: number analyzed (Participants) | 13
  Change from Baseline at Day 7 | -4.42 (2.964)

7. Secondary Outcome: Change From Baseline in the TETRAS Upper Limb Individual Items (Performance Subscale Items 4a, 4b, or 4c) Scores at Day 7
Description: The TETRAS individual item score is the sum of the TETRAS Performance Subscale items 4a, 4b, or 4c scores [4a: forward outstretched postural tremor (FOPT), 4b: lateral "wing beating" postural tremor (LWBPT), 4c: kinetic tremor] from both sides of the body. Each TETRAS score ranges from 0 to 4; the total score ranges from 0 to 16; higher scores indicate more severe tremor. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) and Day 7 (8 hours postdose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: SAGE-217 Capsules
Number analyzed (Participants) | 14
score on a scale
  FOPT at Baseline (Day 1) | 4.14 (0.989)
  Change from Baseline in FOPT at Day 7: number analyzed (Participants) | 13
  Change from Baseline in FOPT at Day 7 | -1.46 (1.070)
  LWBPT at Baseline (Day 1) | 4.18 (0.932)
  Change from Baseline in LWBPT at Day 7: number analyzed (Participants) | 13
  Change from Baseline in LWBPT at Day 7 | -1.31 (1.011)
  Kinetic Tremor at Baseline (Day 1) | 4.54 (0.720)
  Change from Baseline in Kinetic Tremor at Day 7 | -1.65 (1.179)

8. Secondary Outcome: Part A: Change From Baseline in TETRAS Performance Subscale Score (Items 6, 7, and 8) at Day 7
Description: The TETRAS Performance Subscale score includes 9 items. Out of these 9 items, Item 6 is Archimedes spirals (AS), Item 7 is Handwriting, and Item 8 is Dot approximation task (DAT). Each item was scored from 0 to 4, for both sides of the body, each item has a total score of 0 to 8, where higher scores indicate more severe tremor. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) and Day 7 (predose)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part A: SAGE-217 Capsules
Number analyzed (Participants) | 14
score on a scale
  AS at Baseline (Day 1) | 4.8 (1.37)
  Change from Baseline in AS at Day 7: number analyzed (Participants) | 13
  Change from Baseline in AS at Day 7 | -1.0 (1.29)
  Handwriting at Baseline (Day 1) | 2.3 (1.07)
  Change from Baseline in Handwriting at Day 7: number analyzed (Participants) | 13
  Change from Baseline in Handwriting at Day 7 | -0.4 (0.77)
  DAT at Baseline (Day 1) | 4.46 (0.692)
  Change from Baseline in DAT at Day 7: number analyzed (Participants) | 13
  Change from Baseline in DAT at Day 7 | -0.96 (0.967)

9. Secondary Outcome: Part B: Change From Randomization in the Kinesia Upper Limb Total Score at Day 14
Description: The accelerometer-based Kinesia upper limb total score is the sum of Kinesia kinetic tremor scores across both sides of the body. The individual items included forward outstretched postural tremor (FOPT), lateral "wing beating" postural tremor (LWBPT), and kinetic tremor (KT) scores from both sides of the body. Each upper limb individual item question score for each side of the body ranges from 0 to 4. The Kinesia upper limb total score ranges from 0 to 24, with higher scores indicating more tremors/greater tremor amplitude. A negative change from Randomization indicates improvement.
Time Frame: Randomization (Day 8, predose) and Day 14 (predose)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: Placebo | Part B: SAGE-217 Capsules
Number analyzed (Participants) | 4 | 4
score on a scale
  Randomization (Day 8) | 7.33 (2.373) | 9.13 (7.236)
  Change from Randomization at Day 14 (predose) | 0.93 (2.380) | 0.55 (0.520)
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: SAGE-217 Capsules; Change from Randomization at Day 14; Test type: Superiority; p = 0.7795, Mixed Model for Repeated Measures (MMRM); Least Squares Mean Difference = -0.38, 95% CI 2-sided [-3.47 to 2.70], Standard Error of Mean 1.326 — Least squares mean difference from Randomization (SAGE-217 - placebo); [other analysis details as in outcome 2, analysis 1]

10. Secondary Outcome: Part B: Change From Randomization in the Kinesia Upper Limb Individual Item Score at Day 14
Description: as for outcome 9
Time Frame: Randomization (Day 8, predose) and Day 14 (predose)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: Placebo | Part B: SAGE-217 Capsules
Number analyzed (Participants) | 4 | 4
score on a scale
  FOPT at Randomization (Day 8) | 1.60 (1.098) | 1.85 (2.983)
  Change from Randomization in FOPT at Day 14 | 0.03 (0.580) | 0.38 (0.591)
  LWBPT at Randomization (Day 8) | 2.40 (0.876) | 3.15 (3.032)
  Change from Randomization in LWBPT at Day 14 | 0.70 (1.553) | 0.03 (0.263)
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: SAGE-217 Capsules; Change from Randomization in Forward outstretched postural tremor (FOPT) at Day 14; Test type: Superiority; p = 0.4846, Mixed Model for Repeated Measures (MMRM); Least Squares Mean Difference = 0.34, 95% CI 2-sided [-0.65 to 1.33], Standard Error of Mean 0.473 — Least squares mean difference from Randomization (SAGE-217 - placebo); [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: SAGE-217 Capsules; Change from Randomization in Lateral "wing beating" postural tremor (LWBPT) at Day 14; Test type: Superiority; p = 0.4567, Mixed Model for Repeated Measures (MMRM); Least Squares Mean Difference = -0.67, 95% CI 2-sided [-2.70 to 1.36], Standard Error of Mean 0.845 — Least squares mean difference from Randomization (SAGE-217 - placebo); [other analysis details as in outcome 2, analysis 1]

11. Secondary Outcome: Part B: Change From Randomization in the TETRAS Upper Limb Total Score at Day 14
Description: The TETRAS performance subscale upper limb total score is the sum of the TETRAS individual item scores from both sides of the body. The TETRAS individual item score included TETRAS Performance Subscale item 4a, 4b and 4c scores [4a: forward outstretched postural tremor (FOPT) and 4b: lateral "wing beating" postural tremor (LWBPT) scores and 4c: Kinetic tremor (KT) score] from both sides of the body. Each individual item score ranges from 0 to 4; The total upper limb score ranges from 0 to 24, higher scores indicate more severe tremor. A negative change from Randomization indicates improvement.
Time Frame: Randomization (Day 8, predose) and Day 14 (predose)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: Placebo | Part B: SAGE-217 Capsules
Number analyzed (Participants) | 4 | 4
score on a scale
  Randomization (Day 8) | 7.88 (1.436) | 7.63 (4.956)
  Change from Randomization at Day 14 | 1.38 (1.109) | 0.63 (0.250)
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: SAGE-217 Capsules; Change from Randomization at Day 14; Test type: Superiority; p = 0.3771, Mixed Model for Repeated Measures (MMRM); Least Squares Mean Difference = -0.76, 95% CI 2-sided [-2.48 to 0.96], Standard Error of Mean 0.850 — Least squares mean difference from Randomization (SAGE-217 - placebo); [other analysis details as in outcome 2, analysis 1]

12. Secondary Outcome: Part B: Change From Randomization in the TETRAS Upper Limb Individual Item (Performance Subscale Items 4a and 4b) Score at Day 14
Description: The TETRAS individual item score is the sum of the TETRAS Performance Subscale item 4a and 4b scores [4a: forward outstretched postural tremor (FOPT) and 4b: lateral "wing beating" postural tremor (LWBPT) scores] from both sides of the body. Each TETRAS score ranges from 0 to 4; the total score ranges from 0 to 16, higher scores indicate more severe tremor. A negative change from Randomization indicates improvement.
Time Frame: Randomization (Day 8, predose) and Day 14 (predose)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: Placebo | Part B: SAGE-217 Capsules
Number analyzed (Participants) | 4 | 4
score on a scale
  FOPT at Randomization (Day 8) | 2.75 (0.500) | 2.63 (1.702)
  Change from Randomization in FOPT at Day 14 | 0.13 (0.629) | 0.00 (0.000)
  LWBPT at Randomization (Day 8) | 2.63 (0.479) | 2.63 (2.056)
  Change from Randomization in LWBPT at Day 14 | 0.38 (0.629) | 0.25 (0.645)
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: SAGE-217 Capsules; Change from Randomization in Forward outstretched postural tremor (FOPT) at Day 14; Test type: Superiority; p = 0.7302, Mixed Model for Repeated Measures (MMRM); Least Squares Mean Difference = -0.14, 95% CI 2-sided [-0.97 to 0.69], Standard Error of Mean 0.415 — Least squares mean difference from Randomization (SAGE-217 - placebo); [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: SAGE-217 Capsules; Change from Randomization in Lateral "wing beating" postural tremor (LWBPT) at Day 14; Test type: Superiority; p = 0.7916, Mixed Model for Repeated Measures (MMRM); Least Squares Mean Difference = -0.13, 95% CI 2-sided [-1.10 to 0.85], Standard Error of Mean 0.467 — Least squares mean difference from Randomization (SAGE-217 - placebo); [other analysis details as in outcome 2, analysis 1]

13. Secondary Outcome: Part B: Change From Randomization in the TETRAS Performance Subscale Item 4c (Kinetic Tremor) Combined Score at Day 14
Description: The TETRAS kinetic tremor combined score is the sum of the TETRAS Performance Subscale item 4c (kinetic tremor) scores from both sides of the body. The TETRAS kinetic tremor score ranges from 0 to 4, the total score for both sides of the body ranges from 0 to 8, higher scores indicate more severe tremor. A negative change from Randomization indicates improvement.
Time Frame: Randomization (Day 8, predose) and Day 14 (predose)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: Placebo | Part B: SAGE-217 Capsules
Number analyzed (Participants) | 4 | 4
score on a scale
  Randomization (Day 8) | 2.50 (0.577) | 2.38 (1.250)
  Change from Randomization at Day 14 | 0.88 (0.479) | 0.38 (0.479)
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: SAGE-217 Capsules; Change from Randomization at Day 14; Test type: Superiority; p = 0.1807, Mixed Model for Repeated Measures (MMRM); Least Squares Mean Difference = -0.47, 95% CI 2-sided [-1.17 to 0.23], Standard Error of Mean 0.340 — Least squares mean difference from Randomization (SAGE-217 - placebo); [other analysis details as in outcome 2, analysis 1]

14. Secondary Outcome: Part B: Change From Baseline in TETRAS Performance Subscale (Items 6, 7, and 8) Score at Day 14
Description: as for outcome 8
Time Frame: Baseline (Day 1) and Day 14 (predose)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part B: Placebo | Part B: SAGE-217 Capsules
Number analyzed (Participants) | 4 | 4
score on a scale
  AS at Baseline (Day 1) | 5.0 (0.82) | 5.3 (1.89)
  Change from Baseline in AS at Day 14 | -1.3 (0.96) | -1.0 (1.15)
  Handwriting at Baseline (Day 1) | 2.3 (0.96) | 3.0 (1.41)
  Change from Baseline in Handwriting at Day 14 | -0.5 (1.00) | -0.5 (0.58)
  DAT at Baseline (Day 1) | 4.63 (0.629) | 4.50 (1.000)
  Change from Baseline in DAT at Day 14 | -1.25 (0.866) | -1.38 (1.250)
Statistical Analysis 1: Comparison: Part B: Placebo vs Part B: SAGE-217 Capsules; Change from Baseline in Archimedes Spirals (AS) at Day 14; Test type: Superiority; p = 0.8709, Mixed Model for Repeated Measures (MMRM); Least Squares Mean Difference = 0.1, 95% CI 2-sided [-1.7 to 1.9], Standard Error of Mean 0.72 — Least squares mean difference from Baseline(SAGE-217 - placebo); [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Part B: Placebo vs Part B: SAGE-217 Capsules; Change from Baseline in Handwriting at Day 14; Test type: Superiority; p = 0.7843, Mixed Model for Repeated Measures (MMRM); Least Squares Mean Difference = -0.2, 95% CI 2-sided [-1.8 to 1.4], Standard Error of Mean 0.65 — Least squares mean difference from Baseline (SAGE-217 - placebo); [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Part B: Placebo vs Part B: SAGE-217 Capsules; Change from Baseline in Dot approximation task (DAT) at Day 14; Test type: Superiority; p = 0.7604, Mixed Model for Repeated Measures (MMRM); Least Squares Mean Difference = -0.31, 95% CI 2-sided [-2.72 to 2.10], Standard Error of Mean 0.984 — Least squares mean difference from Baseline (SAGE-217 - placebo; [other analysis details as in outcome 2, analysis 1]

15. Secondary Outcome: Part C: Change From Baseline in the Kinesia Upper Limb Individual Item Score at Day 15
Description: as for outcome 4
Time Frame: Baseline (Day 1) and Day 15
Population: The Efficacy Population consisted of all participants who completed at least 1 dose of study drug in the capsule formulation in Part C and had at least 1 postdose efficacy evaluation. Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part C: SAGE-217 Capsules
Number analyzed (Participants) | 16
score on a scale
  FOPT at Baseline (Day 1) | 2.98 (1.626)
  Change from Baseline in FOPT at Day 15: number analyzed (Participants) | 13
  Change from Baseline in FOPT at Day 15 | -0.53 (1.156)
  LWBPT at Baseline (Day 1) | 4.41 (1.548)
  Change from Baseline in LWBPT at Day 15: number analyzed (Participants) | 12
  Change from Baseline in LWBPT at Day 15 | -0.93 (1.497)
  Kinetic tremor at Baseline (Day 1) | 4.28 (1.275)
  Change from Baseline in Kinetic tremor at Day 15: number analyzed (Participants) | 13
  Change from Baseline in Kinetic tremor at Day 15 | -0.51 (1.229)
Statistical Analysis 1: Comparison: Part C: SAGE-217 Capsules; Change from Baseline in Forward outstretched postural tremor (FOPT) at Day 15; Test type: Other; p = 0.1333, Mixed Model for Repeated Measures (MMRM); Least Squares Mean Difference = -0.48, 95% CI 2-sided [-1.13 to 0.17], Standard Error of Mean 0.301 — Least squares mean difference from Baseline (SAGE-217); [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Part C: SAGE-217 Capsules; Change from Baseline in Lateral "wing beating" postural tremor (LWBPT) at Day 15; Test type: Other; p = 0.0572, Mixed Model for Repeated Measures (MMRM); Least Squares Mean Difference = -0.81, 95% CI 2-sided [-1.64 to 0.03], Standard Error of Mean 0.389 — Least squares mean difference from Baseline (SAGE-217); [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Part C: SAGE-217 Capsules; Change from Baseline in Kinetic tremor (KT) at Day 15; Test type: Other; p = 0.0707, Mixed Model for Repeated Measures (MMRM); Least Squares Mean Difference = -0.50, 95% CI 2-sided [-1.05 to 0.05], Standard Error of Mean 0.255 — Least squares mean difference from Baseline (SAGE-217); [other analysis details as in outcome 2, analysis 1]

16. Secondary Outcome: Part C: Change From Baseline in the TETRAS Upper Limb Total Score at Day 15
Description: The TETRAS performance subscale upper limb total score is the sum of the TETRAS individual item scores from both sides of the body. Each individual item score ranges from 0 to 4; The total upper limb score ranges from 0 to 24, higher scores indicate more severe tremor. A negative change indicates improvement.
Time Frame: Baseline (Day 1) and Day 15
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part C: SAGE-217 Capsules
Number analyzed (Participants) | 17
score on a scale
  Baseline (Day 1) | 12.82 (1.952)
  Change from Baseline at Day 15: number analyzed (Participants) | 15
  Change from Baseline at Day 15 | -1.60 (2.436)
Statistical Analysis 1: Comparison: Part C: SAGE-217 Capsules; Change from Baseline at Day 15; Test type: Other; p = 0.0278, Mixed Model for Repeated Measures (MMRM); Least Squares Mean Difference = -1.53, 95% CI 2-sided [-2.87 to -0.19], Standard Error of Mean 0.628 — Least squares mean difference from Baseline (SAGE-217); [other analysis details as in outcome 2, analysis 1]

17. Secondary Outcome: Part C: Change From Baseline in the TETRAS Upper Limb Individual Item (Performance Subscale Items 4a and 4b) Score at Day 15
Description: The TETRAS individual item score is the sum of the TETRAS Performance Subscale item 4a and 4b scores [4a: forward outstretched postural tremor (FOPT) and 4b: lateral "wing beating" postural tremor (LWBPT) scores] from both sides of the body. Each TETRAS score ranges from 0 to 4; the total score ranges from 0 to 16, higher scores indicate more severe tremor. A negative change from Baseline indicates improvement.
Time Frame: Baseline (Day 1) and Day 15
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part C: SAGE-217 Capsules
Number analyzed (Participants) | 17
score on a scale
  FOPT at Baseline (Day 1) | 3.79 (0.867)
  Change from Baseline in FOPT at Day 15: number analyzed (Participants) | 15
  Change from Baseline in FOPT at Day 15 | -0.13 (1.060)
  LWBPT at Baseline (Day 1) | 4.47 (0.695)
  Change from Baseline in LWBPT at Day 15: number analyzed (Participants) | 15
  Change from Baseline in LWBPT at Day 15 | -0.80 (0.902)
  Kinetic tremor at Baseline (Day 1) | 4.56 (0.726)
  Change from Baseline in Kinetic tremor at Day 15: number analyzed (Participants) | 15
  Change from Baseline in Kinetic tremor at Day 15 | -0.67 (0.838)
Statistical Analysis 1: Comparison: Part C: SAGE-217 Capsules; Change from Baseline in Forward outstretched postural tremor (FOPT) at Day 15; Test type: Other; p = 0.9579, Mixed Model for Repeated Measures (MMRM); Least Squares Mean Difference = -0.01, 95% CI 2-sided [-0.57 to 0.54], Standard Error of Mean 0.258 — Least squares mean difference from Baseline (SAGE-217); [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Part C: SAGE-217 Capsules; Change from Baseline in Lateral "wing beating" postural tremor (LWBPT) at Day 15; Test type: Other; p = 0.0039, Mixed Model for Repeated Measures (MMRM); Least Squares Mean Difference = -0.80, 95% CI 2-sided [-1.31 to -0.30], Standard Error of Mean 0.234 — Least squares mean difference from Baseline (SAGE-217); [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Part C: SAGE-217 Capsules; Change from Baseline in Kinetic tremor (KT) at Day 15; Test type: Other; p = 0.0099, Mixed Model for Repeated Measures (MMRM); Least Squares Mean Difference = -0.67, 95% CI 2-sided [-1.14 to -0.19], Standard Error of Mean 0.223 — Least squares mean difference from Baseline (SAGE-217); [other analysis details as in outcome 2, analysis 1]

18. Secondary Outcome: Part C: Change From Baseline in TETRAS Performance Subscale (Items 6, 7, and 8) Scores at Day 15
Description: as for outcome 8
Time Frame: Baseline (Day 1) and Day 15
Population: as for outcome 15
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part C: SAGE-217 Capsules
Number analyzed (Participants) | 17
score on a scale
  AS at Baseline (Day 1): number analyzed (Participants) | 16
  AS at Baseline (Day 1) | 4.5 (1.97)
  Change from Baseline in AS at Day 15: number analyzed (Participants) | 14
  Change from Baseline in AS at Day 15 | -0.6 (1.55)
  Handwriting at Baseline (Day 1) | 2.4 (1.06)
  Change from Baseline in Handwriting at Day 15: number analyzed (Participants) | 15
  Change from Baseline in Handwriting at Day 15 | -0.5 (0.74)
  DAT at Baseline (Day 1) | 4.25 (0.640)
  Change from Baseline in DAT at Day 15: number analyzed (Participants) | 15
  Change from Baseline in DAT at Day 15 | -0.23 (0.594)
Statistical Analysis 1: Comparison: Part C: SAGE-217 Capsules; Change from Baseline in Archimedes spirals (AS) at Day 15; Test type: Other; p = 0.1595, Mixed Model for Repeated Measures (MMRM); Least Squares Mean Difference = -0.6, 95% CI 2-sided [-1.5 to 0.3], Standard Error of Mean 0.41 — Least squares mean difference from Baseline (SAGE-217); [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 2: Comparison: Part C: SAGE-217 Capsules; Change from Baseline in Handwriting at Day 15; Test type: Other; p = 0.0126, Mixed Model for Repeated Measures (MMRM); Least Squares Mean Difference = -0.5, 95% CI 2-sided [-0.9 to -0.1], Standard Error of Mean 0.19 — Least squares mean difference from Baseline (SAGE-217); [other analysis details as in outcome 2, analysis 1]
Statistical Analysis 3: Comparison: Part C: SAGE-217 Capsules; Change from Baseline in Dot approximation task (DAT) at Day 15; Test type: Other; p = 0.1536, Mixed Model for Repeated Measures (MMRM); Least Squares Mean Difference = -0.23, 95% CI 2-sided [-0.55 to 0.10], Standard Error of Mean 0.151 — Least squares mean difference from Baseline (SAGE-217); [other analysis details as in outcome 2, analysis 1]

19. Secondary Outcome: Parts A, B and C: Number of Participants With at Least One Treatment-Emergent Adverse Event (TEAE) or Serious Adverse Event (SAE)
Description: An Adverse Event (AE) was defined as any untoward medical occurrence associated with the use of a drug in humans, whether or not considered drug-related. Adverse events that occurred after the first administration of study drug were denoted as TEAEs. A Serious Adverse Event (SAE) was an AE occurring during any study phase and at any dose of the study drug, comparator, or placebo, that fulfilled the following outcomes: death, a life-threatening adverse event, inpatient hospitalization or prolongation of existing hospitalization, a persistent or significant incapacity or substantial disruption of the ability to conduct normal functions, or a congenital anomaly/birth defect. Important medical events that may not result in death, be life-threatening, or require hospitalization may be considered serious when, based upon appropriate medical judgment, they may jeopardize the participant and may require medical or surgical intervention to prevent one of the outcomes listed in this definition.
Time Frame: From first dose of study drug through 14 days after the last dose (Up to 28 days)
Population: The Safety Population consisted of all participants who were administered at least 1 dose of open-label study drug (Parts A and C) or double-blind study drug (Part B).
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: SAGE-217 Oral Solution | Part A: SAGE-217 Capsules | Part B: Placebo | Part B: SAGE-217 Capsules | Part C: SAGE-217 Capsules
Number analyzed (Participants) | 2 | 14 | 4 | 4 | 18
Participants
  At Least One TEAE | 2 | 7 | 0 | 1 | 10
  SAE | 1 | 0 | 0 | 0 | 0

20. Secondary Outcome: Part A, B and C: Number of Participants With Suicidal Ideation as Assessed by the Columbia-Suicide Severity Rating Scale (C-SSRS) Score
Description: The C-SSRS consists of a baseline and post-baseline (PB) evaluation that assesses the lifetime experience of the participants with suicidal ideation and behavior. The data for suicidal ideation were summarized for participants who answered 'Yes'. Suicide ideation was categorized as 1) wish to be dead and 2) non-specific active suicidal thoughts.
Time Frame: Baseline and post-baseline (up to 28 days)
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Groups:
- Part A: SAGE-217 Oral Solution: Participants received SAGE-217 10 mg on Day 1, 20 mg on Day 2 and 30 mg on Days 3 to 7 as an oral solution with food in the morning.
- Part A: SAGE-217 Capsules: Participants in Part A received a 10-mg dose of SAGE-217, capsules administered with food in the morning on Day 1, 20 mg with food on Day 2 and 30 mg with food daily on Days 3 to 7.
- Part C: SAGE-217 Capsules: Participants received a 10-mg dose of SAGE-217 administered with food in the evening on Day 1, 20 mg with food in the evening on Day 2, and 30 mg with food in the evening on Day 3. From Day 4 through 14 participants received a total 40-mg daily dose with food in the evening.
Arm/Group | Part A: SAGE-217 Oral Solution | Part A: SAGE-217 Capsules | Part B: Placebo | Part B: SAGE-217 Capsules | Part C: SAGE-217 Capsules
Number analyzed (Participants) | 2 | 14 | 4 | 4 | 18
Participants
  Wish to be Dead (baseline) | 0 | 0 | 1 | 0 | 0
  Wish to be Dead (PB) | 0 | 0 | 1 | 0 | 0
  Non-Specific Active Suicidal Thoughts (baseline) | 0 | 0 | 0 | 0 | 0
  Non-Specific Active Suicidal Thoughts (PB) | 0 | 0 | 0 | 0 | 0

21. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs
Description: Vital signs included heart rate, respiratory rate, temperature, and blood pressure.
Time Frame: Up to 28 days
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: SAGE-217 Oral Solution | Part A: SAGE-217 Capsules | Part B: Placebo | Part B: SAGE-217 Capsules | Part C: SAGE-217 Capsules
Number analyzed (Participants) | 2 | 14 | 4 | 4 | 18
Participants | 0 | 0 | 0 | 0 | 0

22. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Parameters
Description: Laboratory parameters included hematology, blood chemistry, and urinalysis.
Time Frame: Up to 28 days
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: SAGE-217 Oral Solution | Part A: SAGE-217 Capsules | Part B: Placebo | Part B: SAGE-217 Capsules | Part C: SAGE-217 Capsules
Number analyzed (Participants) | 2 | 14 | 4 | 4 | 18
Participants | 0 | 0 | 0 | 0 | 0

23. Secondary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Values
Description: A 12-lead ECG was performed.
Time Frame: Up to 28 days
Population: as for outcome 19
Measure: Count of Participants; unit: Participants
Arm/Group | Part A: SAGE-217 Oral Solution | Part A: SAGE-217 Capsules | Part B: Placebo | Part B: SAGE-217 Capsules | Part C: SAGE-217 Capsules
Number analyzed (Participants) | 2 | 14 | 4 | 4 | 18
Participants | 0 | 0 | 0 | 0 | 0

24. Secondary Outcome: Parts A and B: Change From Baseline in Stanford Sleepiness Scale (SSS)
Description: The SSS was designed to quickly assess how alert a subject is feeling. Degrees of sleepiness and alertness are rated on a scale of 1 to 7, where the lowest score of 1 indicates the subject is "feeling active, vital, alert, or wide awake" and the highest score of 7 indicates the participant is "no longer fighting sleep, sleep onset soon; having dream-like thoughts". Greater changes from baseline indicate greater sedation. A positive change from baseline indicates improvement.
Time Frame: Baseline (Day 1), Day 7 (predose) for Part A, Day 14 (predose) for Part B
Population: The Safety Population consisted of all participants who were administered at least 1 dose of open-label study drug (Parts A and C) or double-blind study drug (Part B). Number analyzed is the number of participants with data available for analysis at the given time point. SSS was not evaluated in Part C.
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Part A: SAGE-217: Participants received a 10-mg dose of SAGE-217, capsules administered with food in the morning on Day 1, 20 mg with food on Day 2 and 30 mg with food daily on Days 3 to 7.
Arm/Group | Part A: SAGE-217 | Part B: Placebo | Part B: SAGE-217 Capsules
Number analyzed (Participants) | 14 | 4 | 4
score on a scale
  Baseline (Day 1) | 2.1 (1.41) | 1.5 (0.58) | 2.3 (1.26)
  Change from Baseline at Day 7 or 14: number analyzed (Participants) | 13 | 4 | 4
  Change from Baseline at Day 7 or 14 | -0.2 (1.42) | -0.5 (0.58) | -0.5 (0.58)

25. Secondary Outcome: Parts A, B and C: Change From Baseline in Bond-Lader Visual Analogue Scale (VAS) Score
Description: Mood was assessed using the Bond-Lader VAS score. This is a 16-part self-administered questionnaire that employs a 100-mm VAS to explore different aspects of self-reported mood. Three factor scores for (alertness, contentedness, and calmness) were calculated using following equations based on normalized VAS scores:
  * Alertness = 0.827X1 + 0.618X3 + 0.755X4 + 0.642X5 + 0.776X6 + 0.635X9 + 0.792X11 + 0.593X12 + 0.614X15;
  * Contentedness = 0.677X7 + 0.697X8 + 0.823X13 + 0.738X14 + 0.594X16; and
  * Calmness = 0.845X2 + 0.677X10,
  where Xi represents a subject's item score after normalization, and i represents the item number from the entire scale (in order from 1-16). A negative change from baseline (CFB) indicated more alertness, more contentedness, and more calmness.
Time Frame: Baseline (Day 1), Day 7 (predose) for Part A, Day 14 (predose) for Part B and Day 15 for Part C
Population: The Safety Population consisted of all participants who were administered at least 1 dose of open-label study drug (Parts A and C) or double-blind study drug (Part B). Number analyzed is the number of participants with data available for analysis at the given time point.
Measure: Mean (Standard Deviation); unit: log(units on a scale)
Arm/Group | Part A: SAGE-217 Capsules | Part B: Placebo | Part B: SAGE-217 Capsules | Part C: SAGE-217 Capsules
Number analyzed (Participants) | 14 | 4 | 4 | 18
log(units on a scale)
  Alertness: Baseline (Day 1) | 18.737 (3.8640) | 18.345 (3.2388) | 21.308 (2.7694) | 18.1248 (4.62487)
  Alertness: CFB at Day 7, 14 or 15: number analyzed (Participants) | 13 | 4 | 4 | 15
  Alertness: CFB at Day 7, 14 or 15 | -0.148 (6.4794) | -2.857 (1.6712) | -1.038 (4.6404) | 1.3095 (5.87702)
  Contentedness: Baseline (Day 1) | 10.281 (2.7813) | 11.284 (0.2150) | 12.545 (1.7398) | 9.8911 (3.53165)
  Contentedness: CFB at Day 7, 14 or 15 | -0.121 (3.1249) | -1.896 (2.2236) | -0.471 (2.5222) | 0.0881 (3.16922)
  Calmness: Baseline (Day 1) | 4.589 (1.2740) | 5.446 (0.7720) | 5.344 (0.7802) | 5.6157 (0.89826)
  Calmness: CFB at Day 7, 14 or 15 | 0.304 (1.4579) | -0.613 (0.4106) | -0.601 (1.4341) | -0.5116 (1.23403)

26. Secondary Outcome: Parts A, B and C: Participant's Feeling After Taking the Study Drug as Assessed by Drug Effects Questionnaire (DEQ-5) Score
Description: Participants responded to 5 DEQs based on how they are feeling after taking the study drug. DEQ-5 were as follows; Q1: Do you FEEL a drug effect right now? Q2: Are you HIGH right now? Q3: Do you DISLIKE any of the effects that you are feeling right now? Q4: Do you LIKE any of the effects that you are feeling right now? Q5: Would you like MORE of the drug you took, right now? The answers were recorded on a 100-mm VAS, with the answer for each being "Not at all" (0 mm) and "Extremely" (100 mm) at the extremes. There were options to record "Not applicable" for questions 3 and 4 if no drug effects were felt and for question 5 prior to administration of study medication, and these participants were excluded from the data summarization. Higher score on Q1 indicates a drug effect; on Q2 indicates feeling high; on Q3 indicates disliking the drug; and on Q4 and Q5 indicates liking the drug.
Time Frame: Baseline (Day 1), Day 7 (2 hours postdose) for Part A, Day 14 (2 hours postdose) for Part B and Day 15 for Part C
Population: as for outcome 25
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Part A: SAGE-217 Capsules | Part B: Placebo | Part B: SAGE-217 Capsules | Part C: SAGE-217 Capsules
Number analyzed (Participants) | 14 | 4 | 4 | 18
units on a scale
  Q1: Day 7, 14 or 15: number analyzed (Participants) | 13 | 4 | 4 | 15
  Q1: Day 7, 14 or 15 | 54.8 (27.56) | 22.5 (18.84) | 33.0 (28.23) | 27.9 (24.57)
  Q2: Day 7, 14 or 15: number analyzed (Participants) | 13 | 4 | 4 | 15
  Q2: Day 7, 14 or 15 | 21.4 (22.56) | 18.0 (21.65) | 24.5 (21.44) | 13.3 (19.72)
  Q3: Day 7, 14 or 15: number analyzed (Participants) | 13 | 4 | 3 | 15
  Q3: Day 7, 14 or 15 | 47.5 (30.63) | 12.0 (7.83) | 46.3 (24.85) | 35.2 (37.04)
  Q4: Day 7, 14 or 15: number analyzed (Participants) | 13 | 4 | 3 | 15
  Q4: Day 7, 14 or 15 | 30.0 (19.65) | 33.5 (32.25) | 33.0 (17.44) | 38.3 (32.48)
  Q5: Day 7, 14 or 15: number analyzed (Participants) | 13 | 4 | 4 | 15
  Q5: Day 7, 14 or 15 | 34.5 (26.13) | 17.8 (18.61) | 23.0 (20.12) | 34.6 (31.11)

ADVERSE EVENTS:
Time Frame: TEAEs were collected from the first dose of study drug through 14 days after the last dose (up to 28 days).
Description: The Safety Population consisted of all participants who were administered at least 1 dose of open-label study drug (Parts A and C) or double-blind study drug (Part B).
Arm/Group | Part A: SAGE-217 Oral Solution | Part A: SAGE-217 Capsules | Part B: Placebo | Part B: SAGE-217 Capsules | Part C: SAGE-217 Capsules
All-Cause Mortality (participants affected / at risk) | 0/2 | 0/14 | 0/4 | 0/4 | 0/18
Serious Adverse Events (participants affected / at risk) | 1/2 | 0/14 | 0/4 | 0/4 | 0/18
Other Adverse Events (participants affected / at risk) | 2/2 | 7/14 | 0/4 | 1/4 | 10/18
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: SAGE-217 Oral Solution (N=2) | Part A: SAGE-217 Capsules (N=14) | Part B: Placebo (N=4) | Part B: SAGE-217 Capsules (N=4) | Part C: SAGE-217 Capsules (N=18)
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part A: SAGE-217 Oral Solution (N=2) | Part A: SAGE-217 Capsules (N=14) | Part B: Placebo (N=4) | Part B: SAGE-217 Capsules (N=4) | Part C: SAGE-217 Capsules (N=18)
Dizziness (Nervous system disorders) | 2 | 3 | 0 | 0 | 4
Somnolence (Nervous system disorders) | 1 | 4 | 0 | 0 | 5
Sedation (Nervous system disorders) | 1 | 2 | 0 | 0 | 2
Amnesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Bradykinesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Muscle contractions involuntary (Nervous system disorders) | 1 | 0 | 0 | 0 | 0
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 0 | 0 | 1
Somnambulism (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Disorientation (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Nervousness (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0
Diplopia (Eye disorders) | 0 | 1 | 0 | 0 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Gastric infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Paraesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 0 | 0 | 1 | 0

LIMITATIONS AND CAVEATS:
Parts A and B were stopped early (in advance of the planned sample size).

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2017-09-05): https://cdn.clinicaltrials.gov/large-docs/81/NCT02978781/Prot_002.pdf
  • Statistical Analysis Plan (2017-12-14): https://cdn.clinicaltrials.gov/large-docs/81/NCT02978781/SAP_000.pdf